CLINICAL TRIAL: NCT03426319
Title: Cardiovascular Status in Patients With Chronic Cortisol Deficiency (Adrenal Insufficiency)
Brief Title: Cardiovascular Status in Adrenal Insufficiency
Acronym: CVCORT-AI
Status: Completed | Type: Observational
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CV-CORT-AI
Record Dates: First submitted 2018-01-08; First posted 2018-02-08 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2018-01

CONDITIONS: Adrenal Insufficiency
Keywords: Primary adrenal insufficiency; Cardiovascular status; Metabolic profile
MeSH Terms: conditions — Adrenal Insufficiency; Addison Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary adrenal insufficiency: Patients with primary adrenal insufficiency on hormone replacement therapy with hydrocortisone.
  Interventions: Diagnostic Test: Cardiovascular evaluation

INTERVENTIONS:
Diagnostic Test: Cardiovascular evaluation — Cardiovascular evaluation includes anamnesis, physical examination, laboratory tests, analysis of endothelial function, 24h blood pressure profile, Holter ECG, echocardiography and cardiac MRI.

SUMMARY:
Within this trial, the cardiovascular status and metabolic profile of patients with chronic primary adrenal insufficiency is evaluated.

DETAILED DESCRIPTION:
An unfavorable metabolic profile in patients with adrenal insufficiency (AI) under hormone replacement therapy with hydrocortisone (HC) has been revealed in one recent analysis. Furthermore an increased cardiovascular (CV) morbidity in AI is assumed. The aim of the study is to evaluate the metabolic profile and cardiovascular status in patients with primary AI. Patients with primary AI under standard replacement therapy with HC undergo detailed CV evaluation (including e.g. laboratory test, analysis of endothelial function, 24h blood pressure profile, Holter ECG, echocardiography and cardiac MRI).

ELIGIBILITY:
Inclusion Criteria:

* Chronic primary adrenal insufficiency
* Adequate hormone replacement therapy (>3 years)
* Age >18 years
* Patient's informed consent

Exclusion Criteria:

* Hormone replacement therapy with an other glucocorticoid than hydrocortisone
* Pharmacotherapy with glucocorticoids
* Congenital adrenal hyperplasia
* Coronary heart disease
* Heart failure
* Systemic disease with (potential) cardiac involvement (e.g. amyloidosis, lung fibrosis)
* Pregnancy
* Chronic alcohol abuse
* Malignant disease
* Arterial hypertension
* Chronic renal failure (MDRD <60)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic primary adrenal insufficiency
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Cardiovascular status - anamnesis | 12 months
  Evaluation of the cardiovascular status of patients with chronic adrenal insufficiency by anamnesis/documentation of cardiovascular risk factors. Prevalence of cardiovascular risk factors (diabetes, hypertension, hyperlipidemia, obesity) in participating patients.
Cardiovascular status - mean systolic blood pressure | 12 months
  Measurement of the systolic resting blood pressure (in mmHg). Analysis of the mean systolic blood pressure (of all participating patients) and the number of patients with increased systolic blood pressure (>140 mmHg).
Cardiovascular status - mean diastolic blood pressure | 12 months
  Measurement of the diastolic resting blood pressure (in mmHg). Analysis of the mean diastolic blood pressure (of all participating patients).
Cardiovascular status - mean BMI | 12 months
  Measurement of weight (in kg) and height (qm); weight and height will be combined to report the Body Mass Index/BMI (kg/qm).
  Analysis of the mean BMI (of all participating patients) and the number of patients with increased BMI (>25 kg/qm).
Cardiovascular status - mean HbA1c | 12 months
  Measurement of HbA1c-values (in %). Analysis of the mean HbA1c-value and the number of patients with increased HbA1c (>6.5%).
Cardiovascular status - mean cholesterol-level | 12 months
  Measurement of cholesterol-levels (in mg/dl). Analysis of the mean cholesterol-level and the number of patients with increased cholesterol-levels (>200mg/dl).
Cardiovascular status - mean triglyceride-level | 12 months
  Measurement of triglyceride-levels (in mg/dl). Analysis of the mean triglyceride-level and the number of patients with increased triglyceride-levels (>200mg/dl).
Cardiovascular status - reactive hyperaemia index | 12 months
  Evaluation of the reactive hyperaemia index (endothelial function). Analysis of the number of patients with a pathological reactive hyperaemia index (pathological results ≤ 1.67).
Cardiovascular status - mean systolic blood pressure (24h blood pressure measurement) | 12 months
  Measurement of the mean systolic blood pressure (in mmHg) by 24h blood pressure profiles. Analysis of the mean systolic blood pressure (of all participating patients) and the number of patients with an increased mean systolic blood pressure (>140 mmHg).
Cardiovascular status - non-dipper-profiles | 12 months
  Documentation of the number of patients with a non-dipper-profile during a 24h blood pressure measurement.
Cardiovascular status - mean ejection fraction | 12 months
  Analysis of the mean ejection fraction (in %) (by echocardiography of all participating patients) and the number of patients with a pathologic ejection fraction (<55%).
Cardiovascular status - diastolic function | 12 months
  Measurement of the diastolic function by echocardiography. Analysis of the number of patients with a pathological diastolic function (E/A ratio; values <1 were rated as pathological).
Cardiovascular status - pathological cardiac MRI | 12 months
  Number of patients with pathological results (ejection fraction (<55%), pericardial effusion, thrombus, adipose tissue, perfusion defects, late enhancement, valvular or wall motion abnormalities).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Wuerzburg, Würzburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bergthorsdottir R, Leonsson-Zachrisson M, Oden A, Johannsson G. Premature mortality in patients with Addison's disease: a population-based study. J Clin Endocrinol Metab. 2006 Dec;91(12):4849-53. doi: 10.1210/jc.2006-0076. Epub 2006 Sep 12. PMID 16968806
- [Background] Erichsen MM, Lovas K, Skinningsrud B, Wolff AB, Undlien DE, Svartberg J, Fougner KJ, Berg TJ, Bollerslev J, Mella B, Carlson JA, Erlich H, Husebye ES. Clinical, immunological, and genetic features of autoimmune primary adrenal insufficiency: observations from a Norwegian registry. J Clin Endocrinol Metab. 2009 Dec;94(12):4882-90. doi: 10.1210/jc.2009-1368. Epub 2009 Oct 26. PMID 19858318
- [Background] Filipsson H, Johannsson G. GH replacement in adults: interactions with other pituitary hormone deficiencies and replacement therapies. Eur J Endocrinol. 2009 Nov;161 Suppl 1:S85-95. doi: 10.1530/EJE-09-0319. Epub 2009 Aug 14. PMID 19684055
- [Background] Johannsson G, Nilsson AG, Bergthorsdottir R, Burman P, Dahlqvist P, Ekman B, Engstrom BE, Olsson T, Ragnarsson O, Ryberg M, Wahlberg J, Biller BM, Monson JP, Stewart PM, Lennernas H, Skrtic S. Improved cortisol exposure-time profile and outcome in patients with adrenal insufficiency: a prospective randomized trial of a novel hydrocortisone dual-release formulation. J Clin Endocrinol Metab. 2012 Feb;97(2):473-81. doi: 10.1210/jc.2011-1926. Epub 2011 Nov 23. PMID 22112807
- [Background] Burger-Stritt S, Pulzer A, Hahner S. Quality of Life and Life Expectancy in Patients with Adrenal Insufficiency: What Is True and What Is Urban Myth? Front Horm Res. 2016;46:171-83. doi: 10.1159/000443918. Epub 2016 May 17. PMID 27211797
- [Background] Stewart PM, Biller BM, Marelli C, Gunnarsson C, Ryan MP, Johannsson G. Exploring Inpatient Hospitalizations and Morbidity in Patients With Adrenal Insufficiency. J Clin Endocrinol Metab. 2016 Dec;101(12):4843-4850. doi: 10.1210/jc.2016-2221. Epub 2016 Sep 13. PMID 27623069